# The Feasibility Study of The Delivery of The Book From Self Help Plus: "Doing What Matters in Times of Stress: An Illustrated Guide"

[NCT ID not yet assigned]

12/11/2020

# **Informed Consent**

### **Informed Consent**

You are kindly invited to participate in the second part of our TÜBİTAK-funded research, called "The Impact of COVID-19 on Mental Health Problems in Turkey and The Feasibility Study of The Delivery of The Book From Self-Help Plus: "Doing What Matters in Times of Stress: An Illustrated Guide" (2020.200.IRB3.080), led by Dr. Ceren Acartürk from the Department of Psychology at Koç University.

### Purpose of the Study and the Procedure

This part of our study is done to evaluate whether you are eligible for the "Feasibility Study of the delivery of the book from Self-Help Plus, "Doing what matters in times of stress: An illustrated guide". At this point, we will be asking you to answer some questions related to the psychological effects of COVID-19. Your participation in the study is entirely voluntary. In case you accept to participate in the study, we will ask you to fill in an online survey, which will take approximately 15 minutes. After assessing your eligibility to receive the intervention, psychologists from our research team will contact you for the five-week-intervention program. During the intervention program, psychologists will make three phone calls (in the beginning, in the middle, and at the end of the program) in total.

### Possible Benefits to the Community and/or Volunteers

Your participation will give us a comprehensive understanding of the psychological problems experienced by people who live in Turkey during COVID-19. Additionally, it will allow us to test the effectiveness of the intervention program developed to address these psychological problems.

### **Confidentiality**

<u>Under any circumstances</u>, the information you provide during the survey will not be matched with your credentials. It will only be used by the research team for academic purposes. The information you give will be kept in an encrypted database in which only the research team may have access. The information you provided will be recycled once the study is completed in an untraceable manner.

### **Participation and Terminating the Study**

Participation in this study is entirely upon your free will, without any coercion or obligation, your voluntary participation is essential. After deciding to participate, you may terminate the study without providing any specific reason at any time.

For your questions and comments, you may contact the responsible researchers: Assoc. Prof. Ceren Acartürk; cacarturk@ku.edu.tr

## Dr. Ersin Uygun; ersinuygun@hotmail.com

I understood the information provided above and my questions are answered to my satisfaction. Without prejudice to my rights to terminate the study at any point, I agree to the conditions specified below and to participate in the study.

- Under any circumstances, the information I provided during the study will not be matched with my identity and will not be shared with anybody outside the research team.
- I agree that the psychologists working with the research team will contact me 3 times via my phone number if I participate in the intervention program.
- I know that my personal information will be recycled in an untraceable manner if my participation in the intervention program is not found eligible.

I agree to participate in the study.

I do not agree to participate in the study.